CLINICAL TRIAL: NCT05625386
Title: Dual-target, High-dose, Transcranial Magnetic Stimulation for Parkinson's Disease With Freezing of Gait
Brief Title: Dual-target, High-dose TMS for PD Patients With FOG
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was halted at the midpoint because the interim analysis demonstrated a large effect size of the DHT group compared with the SCT group (Cohen's d = 1.58).
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, WANG KAI, Head, Dept of Neurology & Medical Psychology, Director, Cognitive Neuropsychology Lab, PRC, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHMU-TMS-FOG-twotargets
Record Dates: First submitted 2022-06-29; First posted 2022-11-22 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2024-04

CONDITIONS: Transcranial Magnetic Stimulation; Freezing of Gait
Keywords: Transcranial Magnetic Stimulation; Freezing of Gait
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dual-target high-dose TMS (DHT) (Experimental): DHT refers to the left primary motor cortex of the lower leg (M1) and dorsolateral prefrontal cortex (DLPFC) receiving 9000 pulses/day of intermittent TBS (iTBS) for 5 consecutive days. Each iTBS sequence in the high-dose stimulation sequence released 900 pulses at a time with a pulse cluster repeated every 200 ms at a frequency of 5 Hz. Each pulse cluster contained three pulses with a frequency of 50 Hz, stimulation time of 2 s, and interval of 8 s. A total of 10 iTBS sessions was performed each day with an interval of 40 min and the daily stimulation dose was 9000 pulses. The order of stimulation for the two targets was randomized across participants and the order of stimulation within participants remained unchanged throughout the session.
  Interventions: Device: transcranial magnetic stimulation
- Dual-target conventional-dose TMS (DCT) (Experimental): DCT refers to the left M1 and DLPFC receiving 1800 pulses/day of iTBS for 5 consecutive days. Each iTBS sequence in the conventional-dose stimulation sequence released 600 pulses at a time with a pulse cluster repeated every 200 ms at a frequency of 5 Hz. Each pulse cluster contained three pulses with a frequency of 50 Hz, stimulation time of 2 s, and interval of 8 s. A total of three iTBS sessions were performed each day with an interval of 40 min and the daily stimulation dose was 1800 pulses.The order of stimulation for the two targets was randomized across participants and the order of stimulation within participants remained unchanged throughout the session.
  Interventions: Device: transcranial magnetic stimulation
- Single-target conventional-dose TMS (SCT) (Active Comparator): SCT refers to the left M1 receiving 1800 pulses/day of iTBS treatment for 5 consecutive days. Each iTBS sequence in the conventional-dose stimulation sequence released 600 pulses at a time with a pulse cluster repeated every 200 ms at a frequency of 5 Hz. Each pulse cluster contained three pulses with a frequency of 50 Hz, stimulation time of 2 s, and interval of 8 s. A total of three iTBS sessions were performed each day with an interval of 40 min and the daily stimulation dose was 1800 pulses.
  Interventions: Device: transcranial magnetic stimulation

INTERVENTIONS:
Device: transcranial magnetic stimulation — TMS was performed using a Magstim Rapid2 transcranial magnetic stimulator (Magstim Company, Whitland, UK) with a 70-mm air-cooled figure-of-eight coil. All stimulations were guided by a frameless neuronavigation system (Brainsight; Rogue Research, Montreal, QC, Canada).

SUMMARY:
The aim of the current study was to verify whether high-dose TMS treatment of the motor and cognitive cortices is more effective in alleviating FOG than conventional-dose TMS of the motor cortex only. Specifically, investigator hypothesized that the effect of dual-target TMS on FOG is better than traditional stimulation of the motor cortex only, and the effect of high-dose TMS is better than conventional doses.

DETAILED DESCRIPTION:
This was an open-label, randomized controlled study. Participants were randomized in a 1:1:1 fashion to receive dual-target, high-dose TMS (DHT), dual-target, conventional-dose TMS (DCT), and single-target, conventional-dose TMS (SCT). SCT was designated as the control group with protocol reference to evidence-based guidelines, while DHT and DCT served as the experimental groups.

DHT refers to the left primary motor cortex of the lower leg (M1) and dorsolateral prefrontal cortex (DLPFC) receiving 9000 pulses/day of intermittent TBS (iTBS) for 5 consecutive days. DCT refers to the left M1 and DLPFC receiving 1800 pulses/day of iTBS for 5 consecutive days. The order of stimulation for the two targets was randomized across participants and the order of stimulation within participants remained unchanged throughout the session. SCT refers to the left M1 receiving 1800 pulses/day of iTBS treatment for 5 consecutive days.

Motor and cognitive measures were performed ("on medication" state) 1 day before TMS (baseline), 1 day after completion of TMS (post), and 1 month after completion of TMS (follow-up). The primary outcome of this study was the change in FOGQ scores from baseline to follow-up. Secondary outcomes included changes in the Unified Parkinson's Disease Rating Scale Part III (UPDRS III), 5 m Timed Up-and-Go test (TUG), FOG-provoking test (Standing-Start 180° Turn Test, SS-180), Stroop color-naming (SCN), Stroop word-reading (SWR), Stroop color-word (SCW), and Color Trails Test interference index (CTTII) from baseline to follow-up.

Evaluate the patient's brain function and structural changes by collecting Rest-EEG，transcranial magnetic stimulation-EEG, near-infrared functional brain imaging (fNIRS）and fMRI.

TMS was performed using a Magstim Rapid2 transcranial magnetic stimulator (Magstim Company, Whitland, UK) with a 70-mm air-cooled figure-of-eight coil. All stimulations were guided by the participant's anatomical image (1 × 1 × 1 mm3) and a frameless neuronavigation system (Brainsight; Rogue Research, Montreal, QC, Canada).

Stimulation intensity: Because each participant had different sensitivity to TMS, the individual Resting Motor Threshold (RMT) was measured before intervention. Specifically, surface electrodes (Ag/AgCl) were attached to both ends of the right abductor pollicis muscle (the ground wire was connected to the ulnar styloid process) and the left finger motor cortex was stimulated one time. The motor-evoked potentials were recorded from the hand muscles. The RMT was considered when the evoked potential > 50 μV occurred in > 5 of 10 consecutive stimulations. The stimulation intensity during intervention was 80% of the RMT in the current study.

Stimulation sequence: Each iTBS sequence in the high-dose stimulation sequence released 900 pulses at a time with a pulse cluster repeated every 200 ms at a frequency of 5 Hz. Each pulse cluster contained three pulses with a frequency of 50 Hz, stimulation time of 2 s, and interval of 8 s. A total of 10 iTBS sessions was performed each day with an interval of 40 min and the daily stimulation dose was 9000 pulses. Each iTBS sequence in the conventional-dose stimulation sequence released 600 pulses at a time with a pulse cluster repeated every 200 ms at a frequency of 5 Hz. Each pulse cluster contained three pulses with a frequency of 50 Hz, stimulation time of 2 s, and interval of 8 s. A total of three iTBS sessions were performed each day with an interval of 40 min and the daily stimulation dose was 1800 pulses.

Stimulation targets: There were two stimulation targets in this study that were used to intervene in the motor and cognitive cortices. The stimulation target of the motor cortex is located in the lower leg of the left primary motor cortex in the Montreal Neurological Institute space (coordinates: -10, -24, 75 [https:/ /afni.nimh.nih.gov/MNI_Atlas]) based on structural MRI. The stimulation target of the cognitive cortex was the left dorsolateral prefrontal cortex, which has the strongest functional connectivity with the executive control network (see Supplementary materials), based on fMRI. Finally, targets were transformed into the native space for each participant by applying an inverse matrix produced during brain structure and function segmentation using SPM12 (www.fil.ion.ucl.ac.uk/spm) and TMStarget software.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of FOG with expertise in movement disorders.
2. the score of item 3 of the FOG questionnaire ≥1.
3. ongoing treatment with a stable dose of any medication for 2 months.
4. 40 years of age or older.

Exclusion Criteria:

1. a history of addiction, psychiatric disorders, or neurological diseases other than PD.
2. focal brain lesions on T1-/T2-weighted fluid-attenuated inversion recovery images.
3. anti-PD medication adjustments during rTMS treatment.
4. history of substance abuse within the past 6 months.
5. nonremovable metal objects in or around the head.
6. previously received rTMS treatment.
7. prior history of seizure or history in first-degree relatives.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2024-02-25 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
The Freezing of Gait Questionnaire (FOGQ) scores | the changes in FOGQ scores from baseline to 1 month after completion of TMS (follow-up).
  This is an very common clinical motor estimating scale for evaluating FOG. 6 items and each item scored between 0 and 4 points (24 scores in total). Higher scores mean a worse outcome

SECONDARY OUTCOMES:
The timed up and go test (TUG) | changes from baseline to 1 month after completion of TMS (follow-up).
  The participants walk for a distance of five meters from a sitting position and come back to the chair after turning 180° around a traffic cone in a 0.7 m × 0.7 m target box .The time during the whole course are measured. The time is recorded in seconds, and the longer the time, the more severe the symptoms.The longer it takes, the worse it gets
Unified Parkinson's Disease Rating Scale III (UPDRSIII) scores | changes from baseline to 1 month after completion of TMS (follow-up).
  This is an very common clinical motor estimating scale, 14 items and 108' in total. Higher scores indicate worse symptoms. Higher scores mean a worse outcome.
Stroop test | changes (SCN, SWR, SCW) from baseline to 1 month after completion of TMS (follow-up).
  stroop color word test is generally divided into three parts: (1) Quick naming of color dot plots (SCN); (2) Recite the nouns representing the color names quickly (SWR); (3) Present a set of cards, in which the nouns representing the color names are written on the cards in different colors, and check the ability of the subjects to distinguish between the color names and the actual colors, as well as the ability to recite the nouns representing the color names quickly (SCW). The degree to which subjects were influenced by font color as an indicator (SCW) of their cognitive control. The longer it takes, the worse it gets.
Color Trails Test interference index (CTTII) | changes rom baseline to 1 month after completion of TMS (follow-up).
  The number color connection test was divided into two parts, A and B. Part A asked the subjects to connect 25 numbers on the paper in order. In Part B, numbers and letters were replaced by numbers of two different colors to eliminate the influence of culture on the test. When the subjects were asked to connect numbers in order, the two graphs were arranged alternately. The measurement index was time, and the longer the time, the more obvious the decline in prompt ability. CTTII=CTT(part B)-CTT(part A). The longer it takes, the worse it gets.
The Standing-Start 180° Turn Test (SS-180) | changes from baseline to 1 month after completion of TMS (follow-up).
  The participants walk for a distance of five meters from a sitting position and come back to the chair after turning 180° around a traffic cone in a 0.7 m × 0.7 m target box.The time during the 180° turn (SS180) are measured. The time is recorded in seconds, and the longer the time, the more severe the symptoms. The longer it takes, the worse it gets.

CONTACTS AND LOCATIONS:
Overall Officials: Kai Wang, Ph.D., Principal Investigator — Anhui Medical University
Locations (1):
- Cognitive Neuropsychology Lab Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No